CLINICAL TRIAL: NCT06694974
Title: A Randomized Controlled Trial for Liver Fibrosis Assessment in Diabetic Patients
Brief Title: Liver Fibrosis Assessment in Diabetic Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 202408147RINA
Record Dates: First submitted 2024-11-07; First posted 2024-11-19 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Type 2 Diabetes; Metabolic Dysfunction-Associated Steatotic Liver Disease
Keywords: Type 2 diabetes patients; metabolic dysfunction-associated steatotic liver disease
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FIB-4 APP group (Experimental)
  Interventions: Behavioral: APP calculation for FIB-4
- standard group (Other)
  Interventions: Behavioral: Standard Care (in control arm)

INTERVENTIONS:
Behavioral: APP calculation for FIB-4 — the investigators plan to use the smartphone App for FIB-4 calculation and notify the patients.
  Arms: FIB-4 APP group
Behavioral: Standard Care (in control arm) — The standard group proceeds as regular practice
  Arms: standard group

SUMMARY:
The investigators plan to use the smartphone App for FIB-4 calculation and increase the awareness of liver fibrosis. These patients might notify and discuss with the physician of their liver fibrosis severity to improve the identification, and management of liver fibrosis. This is to establish a patient-centered clinical pathway to identify patients with advanced fibrosis in type 2 diabetes patients. The investigators plan to conduct this randomized controlled trial of two groups: FIB-4 APP group and the standard care group. The primary end point is the referral rate of patients with advanced fibrosis (FIB-4 ≥ 2.67).

DETAILED DESCRIPTION:
Non-alcoholic fatty liver disease (NAFLD) is the most common form of chronic liver disease in people with type 2 diabetes. Patients with prediabetes/type 2 diabetes or 2 or more metabolic risk factors are at higher risk for hepatic fibrosis. Type 2 diabetes increases the risk of cirrhosis, cirrhotic complications and liver-related mortality. According to the American Gastroenterology Association guideline, NAFLD screening should be considered for individuals older than 40 years with type 2 diabetes mellitus.

The American diabetes association now advises screening all adults with type 2 diabetes or prediabetes, particularly those with obesity or cardiometabolic risk factors or established cardiovascular disease for clinically significant liver fibrosis (defined as moderate fibrosis to cirrhosis) using a calculated fibrosis-4 index (FIB-4), even those with normal liver enzyme levels.4 People with type 1 diabetes who have obesity, hepatic steatosis, or elevated aminotransferases should also screen for NAFLD. The recommended screening tool is the fibrosis-4 index (FIB-4), a calculation that includes the patient's age, liver enzyme levels, and platelet counts. A score of 1.3 or higher is considered high risk for clinically significant fibrosis, and above 2.67 is very high-risk.

According to a recent study of 1918 patients who received screening Fibroscan, 72.8% had steatosis, and 17.1% had advanced fibrosis (Fibroscan >= 9.6kpa). In another study in Malaysia, among 557 type 2 DM patients who received Fibroscan, 72.4% had NAFLD, and 21% had advanced fibrosis(Fibroscan >= 9.6kpa). Another study screened 561 type 2 diabetes patients in the US, 70% had steatosis, and 9% had advanced fibrosis (Fibroscan >= 9.7kpa). Overall, the prevalence of steatotic liver disease is 70%, and the percentage of advanced fibrosis (>=F3) is 9-21%.

However, the screening of NAFLD in type 2 diabetes patients are underutilized. Because there is still a significant knowledge gap in the clinicians for the identification, diagnosis, and management of NAFLD. There is no country had a national or subnational strategy for NAFLD. Several clinical pathways to facilitate the evaluation of NAFLD in type 2 diabetes patients are developing now. Instead of relying on active assessment by clinicians, automated fibrosis score calculation using the FIB-4 index followed by reminder messages in the electronic clinical management system increased appropriate referral for hepatology assessment or further fibrosis tests in patients with increased fibrosis scores from 3.1% to 33.3%. However, there is still more than 2/3 of patients was not referred for further fibrosis evaluation.

The electronic notification system is not widely available for all clinics, while nearly every patient has the mobile phone. Applying the notification system through the smartphone APP is beneficial for the patients to participate actively for their personal health management and improving disease awareness.

The investigators plan to use the smartphone App for FIB-4 calculation and increase the awareness of liver fibrosis. These patients might notify and discuss with the physician of their liver fibrosis severity to improve the identification, and management of liver fibrosis. This is to establish a patient-centered clinical pathway to identify patients with advanced fibrosis in type 2 diabetes patients. The investigators plan to conduct this randomized controlled trial of two groups: FIB-4 APP group and the standard care group. The primary end point is the referral rate of patients with advanced fibrosis (FIB-4 ≥ 2.67).

ELIGIBILITY:
Inclusion Criteria:

1. Type 2 diabetes patients, regular follow-up in OPD every 3 months
2. Age 35-65 (Because FIB-4 is not accurate in people with age <35 or > 65)

Exclusion Criteria:

1. Patients are regularly follow the investigators at the liver clinic for liver disease
2. Active malignancy
3. Hematology disease with thrombocytopenia
4. Pregnant patients with type 2 diabetes

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 540 (Estimated)
Dates: Start 2024-11-22 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The hepatology clinic referral rate if FIB-4 ≥ 2.67 (advanced fibrosis, F3) | through study completion, an average of 1 year
  Number of patients with FIB-4 ≥ 2.67 being referred to hepatology clinic, divided by total number of patients with FIB-4 ≥ 2.67.

SECONDARY OUTCOMES:
The percentage of patients examined by Fibroscan in each group with FIB4≥2.67 | through study completion, an average of 1 year
  The number of patients with a FIB-4 ≥ 2.67 and received the fibroscan test, divided by the total number of patients with a FIB-4 ≥ 2.67
The hepatology clinic referral rate if FIB-4 ≥ 1.3 and <2.67 in individual groups | through study completion, an average of 1 year
  The number of patients with FIB-4 ≥ 1.3 and <2.67 and referred to the hepatology clinic, divided by the total number of patients with FIB-4 ≥ 1.3 and <2.67
Incidence rate of liver cirrhosis in individual groups | through study completion, an average of 1 year
  Patients diagnosed with liver cirrhosis clinically, divided by the total number of patients in the individual group
The hepatology clinic referral rate of patients with FIB-4 <1.3 in individual groups | through study completion, an average of 1 year
  The number of patients with FIB-4 <1.3 and referred to hepatology clinic, divided by the total number of patients with FIB-4 <1.3

CONTACTS AND LOCATIONS:
Overall Officials: Tung Hung Su, MD, PhD, Principal Investigator — Department of Internal Medicine
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
To protect the patients' privacy information.

REFERENCES:
- [Background] Zhang X, Yip TC, Wong GL, Leow WX, Liang LY, Lim LL, Li G, Ibrahim L, Lin H, Lai JCT, Chim AM, Chan HLY, Kong AP, Chan WK, Wong VW. Clinical care pathway to detect advanced liver disease in patients with type 2 diabetes through automated fibrosis score calculation and electronic reminder messages: a randomised controlled trial. Gut. 2023 Nov 24;72(12):2364-2371. doi: 10.1136/gutjnl-2023-330269. PMID 37549979
- [Background] Lazarus JV, Mark HE, Villota-Rivas M, Palayew A, Carrieri P, Colombo M, Ekstedt M, Esmat G, George J, Marchesini G, Novak K, Ocama P, Ratziu V, Razavi H, Romero-Gomez M, Silva M, Spearman CW, Tacke F, Tsochatzis EA, Yilmaz Y, Younossi ZM, Wong VW, Zelber-Sagi S, Cortez-Pinto H, Anstee QM; NAFLD policy review collaborators. The global NAFLD policy review and preparedness index: Are countries ready to address this silent public health challenge? J Hepatol. 2022 Apr;76(4):771-780. doi: 10.1016/j.jhep.2021.10.025. Epub 2021 Dec 9. PMID 34895743
- [Background] Younossi ZM, Ong JP, Takahashi H, Yilmaz Y, Eguc Hi Y, El Kassas M, Buti M, Diago M, Zheng MH, Fan JG, Yu ML, Wai-Sun Wong V, Alswat K, Chan WK, Mendez-Sanchez N, Burra P, Bugianesi E, Duseja AK, George J, Papatheodoridis GV, Saeed H, Castera L, Arrese M, Kugelmas M, Romero-Gomez M, Alqahtani S, Ziayee M, Lam B, Younossi I, Racila A, Henry L, Stepanova M; Global Nonalcoholic Steatohepatitis Council. A Global Survey of Physicians Knowledge About Nonalcoholic Fatty Liver Disease. Clin Gastroenterol Hepatol. 2022 Jun;20(6):e1456-e1468. doi: 10.1016/j.cgh.2021.06.048. Epub 2021 Jul 3. PMID 34229038
- [Background] Lomonaco R, Godinez Leiva E, Bril F, Shrestha S, Mansour L, Budd J, Portillo Romero J, Schmidt S, Chang KL, Samraj G, Malaty J, Huber K, Bedossa P, Kalavalapalli S, Marte J, Barb D, Poulton D, Fanous N, Cusi K. Advanced Liver Fibrosis Is Common in Patients With Type 2 Diabetes Followed in the Outpatient Setting: The Need for Systematic Screening. Diabetes Care. 2021 Feb;44(2):399-406. doi: 10.2337/dc20-1997. Epub 2020 Dec 21. PMID 33355256
- [Background] Lai LL, Wan Yusoff WNI, Vethakkan SR, Nik Mustapha NR, Mahadeva S, Chan WK. Screening for non-alcoholic fatty liver disease in patients with type 2 diabetes mellitus using transient elastography. J Gastroenterol Hepatol. 2019 Aug;34(8):1396-1403. doi: 10.1111/jgh.14577. Epub 2019 Jan 21. PMID 30551263
- [Background] Kwok R, Choi KC, Wong GL, Zhang Y, Chan HL, Luk AO, Shu SS, Chan AW, Yeung MW, Chan JC, Kong AP, Wong VW. Screening diabetic patients for non-alcoholic fatty liver disease with controlled attenuation parameter and liver stiffness measurements: a prospective cohort study. Gut. 2016 Aug;65(8):1359-68. doi: 10.1136/gutjnl-2015-309265. Epub 2015 Apr 14. PMID 25873639
- [Background] American Diabetes Association Professional Practice Committee. 4. Comprehensive Medical Evaluation and Assessment of Comorbidities: Standards of Care in Diabetes-2024. Diabetes Care. 2024 Jan 1;47(Suppl 1):S52-S76. doi: 10.2337/dc24-S004. PMID 38078591
- [Background] Long MT, Noureddin M, Lim JK. AGA Clinical Practice Update: Diagnosis and Management of Nonalcoholic Fatty Liver Disease in Lean Individuals: Expert Review. Gastroenterology. 2022 Sep;163(3):764-774.e1. doi: 10.1053/j.gastro.2022.06.023. Epub 2022 Jul 14. PMID 35842345
- [Background] Castera L, Cusi K. Diabetes and cirrhosis: Current concepts on diagnosis and management. Hepatology. 2023 Jun 1;77(6):2128-2146. doi: 10.1097/HEP.0000000000000263. Epub 2023 Jan 13. PMID 36631005
- [Background] Wattacheril JJ, Abdelmalek MF, Lim JK, Sanyal AJ. AGA Clinical Practice Update on the Role of Noninvasive Biomarkers in the Evaluation and Management of Nonalcoholic Fatty Liver Disease: Expert Review. Gastroenterology. 2023 Oct;165(4):1080-1088. doi: 10.1053/j.gastro.2023.06.013. Epub 2023 Aug 4. PMID 37542503
- See also: Related Info — https://reg.ntuh.gov.tw/RECManageSystem/